CLINICAL TRIAL: NCT07152015
Title: Examination of Sarcopenia and Respiratory Functions in Multiple Sclerosis
Brief Title: Multiple Sclerosis, Sarcopenia and Respiration
Status: Not yet recruiting | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, tuba kolaylı, Lecturer, Uskudar University
Other Study IDs: sar123
Record Dates: First submitted 2025-08-18; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; sarcopenia; inspiratory muscle strength
MeSH Terms: conditions — Multiple Sclerosis; Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sarcopenic MS
- Nonsarcopenic MS

SUMMARY:
The goal of this observational study is to evaluate the relationship between respiratory function and sarcopenia in people with multiple sclerosis.

The main questions it aims to answer are:

Is there a relationship between muscle structure and respiratory muscle strength/pulmonary function in MS patients?

Undergo a single session of respiratory muscle strength measurement (e.g., maximal inspiratory pressure [MIP], maximal expiratory pressure [MEP]) Perform spirometry to assess pulmonary function

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with MS by a neurologist
* Being diagnosed with Sarcopenia
* No history of attacks in the last 3 months
* Able to walk with and without support (EDSS<6.5)

Exclusion Criteria:

* Having concomitant lung and heart disease
* Mini Mental score below 24
* Being in pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient with Multiple Sclerosis Disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity | 1 day (The evaluation will be done one-time)
  FVC, defined as the total volume of air that can be forcibly exhaled after full inspiration, will be recorded with spirometry using the Cosmed Pony FX device, following ATS guidelines.
Forced Expiratory Volume in 1 second (FEV1) | 1 day (The evaluation will be done one-time)
  FEV1, spirometric evaluation of the maximum volume of air exhaled in the first second of a forced breath, will be measured using the Cosmed Pony FX device (Rome, Italy) in accordance with ATS standards.
FEV1/FVC Ratio (%) | 1 day (The evaluation will be done one-time)
  The ratio of FEV1 to FVC (FEV1/FVC) will be obtained as an index of airflow limitation. This ratio will be calculated from spirometry values measured with the Cosmed Pony FX device under ATS standards.
Maximal Inspiratory Pressure | 1 day (The evaluation will be done one-time)
  MIP, reflecting inspiratory muscle strength, will be assessed through maximal inspiratory efforts against a closed airway, using the Cosmed Pony FX device according to ATS recommendations.
Maximal Expiratory Pressure | 1 day (The evaluation will be done one-time)
  MEP, representing expiratory muscle strength, will be determined by maximal expiratory efforts against a closed airway. Measurements will be obtained with the Cosmed Pony FX device (Rome, Italy) according to ATS standards

SECONDARY OUTCOMES:
and grip strength measurement | 1 day (The evaluation will be done one-time)
  Muscle strength assessment will do by measuring handgrip strength. The measurement is performed with the JAMAR hand dynamometer upon the recommendation of the American Hand Therapists Association.
Skeletal Muscle Index (SMI, kg/m²) | 1 day (The evaluation will be done one-time)
  Skeletal Muscle Index (SMI) will be assessed using bioelectrical impedance analysis (BIA). SMI will be calculated as appendicular skeletal muscle mass (kg) divided by height squared (m²). Measurements will be performed once at baseline under standard BIA testing conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Kolaylı Çerezci, PhD(c), Principal Investigator — Uskudar University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sawaya Y, Shiba T, Ishizaka M, Hirose T, Sato R, Kubo A, Urano T. Sarcopenia is not associated with inspiratory muscle strength but with expiratory muscle strength among older adults requiring long-term care/support. PeerJ. 2022 Feb 17;10:e12958. doi: 10.7717/peerj.12958. eCollection 2022. PMID 35194529